CLINICAL TRIAL: NCT03859726
Title: Predictive Value of Sublingual Microcirculation and Peripheral Tissue Oxygen Monitoring in Sepsis Patients With Successful Fluid Resuscitation
Brief Title: Predictive Value of Sublingual Microcirculation and Peripheral Tissue Oxygen Monitoring
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 201902035
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2019-01

CONDITIONS: Sepsis
Keywords: Sepsis, NIRS, sublingual microcirculation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Compliance group: 6hLC≥10% NIRS Sublingual microcirculation
  Interventions: Diagnostic Test: NIRS; Diagnostic Test: Sublingual microcirculation
- Non compliance group: 6hLC<10%

INTERVENTIONS:
Diagnostic Test: NIRS — Near-infrared spectroscopy (NIRS) offers non-invasive, in-vivo, real-time monitoring of tissue oxygenation. Changes in regional tissue oxygenation as detected by NIRS may reflect the delicate balance between oxygen delivery and consumption.
  Groups: Compliance group
Diagnostic Test: Sublingual microcirculation — The sidestream dark field (SDF) imaging devices provide high contrast images of the microvasculature.
  Groups: Compliance group

SUMMARY:
Change and predictive Value of Sublingual Microcirculation and Peripheral Tissue Oxygen Monitoring in Sepsis Patients With Successful Fluid Resuscitation

DETAILED DESCRIPTION:
Fluid therapy for sepsis patients has always been a research hotspot. Early studies suggest that early goal-directed therapy (EGDT) can reduce mortality in patients with sepsis and septic shock, which is included in the guidelines. However, recent studies suggest that EGDT does not reduce mortality. This may be related to the fact that EGDT only pays attention to systemic circulation and neglects microcirculation.

In the past few decades, arterial blood pressure, blood lactic acid and other circulatory indicators have been the target of septic shock treatment, but normal systemic circulation does not mean normal tissue perfusion. Obstacles to tissue perfusion, oxygenation and microcirculation may still exist. At the same time, compared with systemic hemodynamic parameters, microcirculation parameters may play a stronger role in predicting the prognosis of sepsis patients. It is believed that the ideal goal of resuscitation therapy for sepsis should be based on whether microcirculation function has been restored or not.

Objective:to observe the success rate of microcirculation imaging and oxygen saturation of peripheral tissues in sepsis patients under the guidance of current guidelines and procedures. At the same time, we compared the predictive value of microcirculation indicators to the prognosis of septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* patients fullfilled the diagnostic criteria of Sepsis 3.0

Exclusion Criteria:

* Patients who were younger than 18 years old，
* pregnant women
* patients who had been admitted to the Intensive Care Unit(ICU for<24 h)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Results for continuous variables with normal distributions were presented as mean±standard deviations (SD)．Results for continuous variables that were not normally distributed were presented as median(Ql，Q1)．
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Sepsis Related Organ Failure Assessment | 72 hours
  SOFA

SECONDARY OUTCOMES:
28-day mortality | 28-day
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang X, Zhang H, Jin R, Li L, Huang L, Wang Z, Peng Q, Ai M, Zhang L. Assessment of Sublingual Microcirculation to Evaluate the Efficacy of Resuscitation Therapy in Septic Shock Patients: A Cohort Study. Shock. 2026 Feb 1;65(2):161-172. doi: 10.1097/SHK.0000000000002708. Epub 2025 Sep 25. PMID 41031817